CLINICAL TRIAL: NCT02728973
Title: Effects of Enhanced Recovery After Surgery (ERAS) Protocol on the Incidence of Postoperative Complications Following Intestinal Surgery
Brief Title: ERAS Protocol on the Incidence of Postoperative Complications Following Intestinal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, Professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: ERASCQ2016
Record Dates: First submitted 2016-03-27; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Complications
Keywords: colorectal resection; enhanced recovery after surgery; Postoperative Complications; length of hospital stay
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ERAS program: The main elements of this program were: preoperative advice, no colon preparation, provision of carbohydrate-rich drinks one day prior and on the morning of surgery, goal directed fluid administration, body temperature control during surgery, avoiding drainages and nasogastric tubes, early mobilization, and the taking of oral fluids in the early postoperative period.
  Interventions: Other: ERAS program
- conventional treatment program: conventional treatment

INTERVENTIONS:
Other: ERAS program — The main elements of this program were: preoperative advice, no colon preparation, provision of carbohydrate-rich drinks one day prior and on the morning of surgery, goal directed fluid administration, body temperature control during surgery, avoiding drainages and nasogastric tubes, early mobilization, and the taking of oral fluids in the early postoperative period.
  Groups: ERAS program

SUMMARY:
Enhanced recovery after surgery (ERAS) was first proposed by Kehlet in Copenhagen Denmark, this is a new concept for the integration of the latest study of the surgical, anesthesia, and nursing. The purpose of optimization measures, reduce patient trauma stress, promote early rehabilitation of patients. The investigators plan to compare the feasibility, clinical effectiveness, and cost savings of an ERAS program with traditional treatment program at a major teaching hospital in China.The investigators will apply ERAS plan or traditional treatment regimens in the treatment of 100 cases of colorectal cancer patients, respectively. And data Compare the two programs about the incidence of postoperative complications, postoperative hospital stay, cost of hospitalization, and readmission rate will be collected.

DETAILED DESCRIPTION:
Major colorectal surgery usually requires a hospital stay of more than 12 days. Inadequate pain management, intestinal dysfunction and immobilisation are the main factors associated with delay in recovery. This study aims to assess the short and medium term results achieved by an enhanced recovery program based on previously published protocols. This prospective study will be performed at a major hospital in China, involved 200 patients. All patients underwent elective colorectal resection for cancer are divided into enhanced recovery program group or conventional treatment group. The main elements of this program were: preoperative advice, no colon preparation, provision of carbohydrate-rich drinks one day prior and on the morning of surgery, goal directed fluid administration, body temperature control during surgery, avoiding drainages and nasogastric tubes, early mobilization, and the taking of oral fluids in the early postoperative period. Perioperative morbidity and mortality data will be collected and the length of hospital stay and protocol compliance recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Elective laparotomy or laparoscopic intestinal surgery.
2. Age ≥ 18 years old.
3. ASA grade II - IV.
4. General anesthesia.

Exclusion Criteria:

1. Patients with cognitive dysfunction and uncooperative subjects.
2. Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receive elective laparotomy or laparoscopic intestinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The difference in postoperative morbidity rate | within postoperative 30 days

SECONDARY OUTCOMES:
length of hospital stay | within postoperative 30 days
mortality | within postoperative 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, MD, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The first Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peng LH, Min S, Jin JY, Wang WJ. Stratified pain management counseling and implementation improving patient satisfaction: a prospective, pilot study. Chin Med J (Engl). 2019 Dec 5;132(23):2812-2819. doi: 10.1097/CM9.0000000000000540. PMID 31856052